CLINICAL TRIAL: NCT05322226
Title: Evaluation of an Addiction Intervention in Candidates for Liver Transplantation
Brief Title: Addiction Intervention in Liver Transplantation Candidates
Acronym: Addictolive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0516
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Transplant; Failure, Liver; Addiction, Alcohol
Keywords: Liver transplantation; Alcohol relapse; Biological markers of alcohol consumption; Addiction follow up
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults undergoing pre- liver transplant assessment (Other): All patients included in the study will have blood and urinary test from their registration on the transplant list and during their classic follow-up with their hepatologist for 12 months to quantify the biological markers of alcoholism (every 3 months). Additional tubes and urine will be collected in order to measure these markers (urinary ethylglucuronide and blood phosphatidylethanol).
  Interventions: Behavioral: Addiction follow-up before and after liver transplantation

INTERVENTIONS:
Behavioral: Addiction follow-up before and after liver transplantation — Addiction consult and follow-up

SUMMARY:
Addiction care is "a la carte treatment", adapted to the motivation and time constrains of users. Thus, various types of psychotherapeutic follow-up can be considered, different addictolytic medications or opioid maintenance therapies can be offered during treatment and hospitalization must be adaptable. In liver transplantation (LT), sustained alcohol relapse is a critical issue because it increases medium and long-term morbidity and mortality. In recent years, the issue of severe acute alcoholic hepatitis as an indication for LT has necessitated increased focus on appropriate alcohol monitoring around liver transplantation. Previously, alcohol consumption in pre- and post-LT period was mainly self-reported. More recently, the biological markers of excessive alcohol consumption have been validated in liver disease and can play a role in liver transplant recipients follow-up.

The investigator hypothesize that standardized targeted addiction monitoring of LT patients decreases the rates of sustained alcohol relapse one year post liver transplantation.

DETAILED DESCRIPTION:
The main objective of this study is to identify the impact of a targeted addiction monitoring of pre- and post-LT patients on rates of sustained alcohol relapse, one year after LT at the Liver Transplant Unit of the University Hospital of Montpellier. The secondary objectives are: (i) to precisely detail all the addiction treatments (medications, psychotherapy types and specific hospitalization) implemented during this follow-up, (ii) to assess the impact of targeted addiction treatment on the tobacco use and other psychoactive substances (PS) consumption rates , (iii) to quantify LT patients' acceptability of referral to addiction-related treatment and care, (iv) to assess the relevance of biological markers of excessive alcohol consumption during pre- and post-LT period.

The investigator will conduct an A'Hern Single-stage Phase II monocentric interventional trial.

All patients undergoing assessment for LT in Montpellier's Liver Transplant Unit will be consecutively included during their first systematic consultation with the addiction specialist. During this interview, the risk of alcohol relapse will be assessed and targeted addiction follow-up will be planned. Starting from the registration on the national waiting list, biological markers of excessive alcohol consumption will be performed every three months and the patient will be referred to the addiction specialist if the results are positive. After LT these evaluations will continue every three months for one year and patients will be referred for addiction treatment as needed. All participants will have a final interview with an addiction specialist one year post LT.

Using the single-stage A'Hern design, a sample size of 65 LT patients is required to distinguish between a maximum futility proportion of 26% of sustained relapses and a minimum efficacy proportion of 13%, with a one-sided significance level of 0,047 and a power of 82,4%. Based on these criteria, the number of patients with sustained relapse must be at least 10 for the proposed treatment to be deemed effective.

Each patient's socio-demographic, medical, hepatological and addiction data will be collected at baseline. All data concerning each patient's targeted addiction follow-ups, biological markers, rates of sustained alcohol relapse, tobacco and PS consumption rates will be noted during the first year after LT.

ELIGIBILITY:
Inclusion Criteria:

* all adults undergoing pre-transplant assessment in the Liver Transplantation Unit of University Hospital of Montpellier, providing oral informed consent.

Exclusion Criteria:

* Patients under protection of justice or unable to receive a clear information.
* Exclusion period determined by previous study
* Pregnent women or breastfeeding
* Patient under guardianship or curatorship
* Not affiliated to french social security

Removal of subjects from study criteria:

* not registered on the liver transplant waiting-list or not transplanted during the study period
* Liver transplantation prior to visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of liver transplant patients with sustained alcohol relapse one year after liver transplant | 1 year
  The rate is defined by at least one positive alcohol marker and a daily amount of alcohol exceeding 3 (women) or 4 (men) drinks per day with the notion of loss of control recorded during addiction interview

SECONDARY OUTCOMES:
Description of addictological means implemented during follow-up. | 1 year
  Addiction physician will choose medications, psychotherapeutic interventions, and hospitalization when appropriate.
  Rate of patients in pre-transplantation evaluated at low risk and with severe relapse at 1 year post liver transplant.
Addiction consult | 1 year
  Rate of patient complying with their appointment
Addiction consult following biology results | 1 year
  Proportion of follow-up addiction consultations having been guided, according to the opinion of the clinician, by the results of the biological markers (and not only by the self-declaration of consumption).
Caracterization of contraindicated patients | 1 year
  Rates and characteristics of patients with temporary and/or permanent addiction contraindication
Rate of transplanted patients with tobacco and other psycoactive substance consumption during the first year after liver transplant | Every 3 months during 1 year
  Smoking cessation is defined declaratively and using an expired CO test (< 6.5 ppm). Psychoactive substance consumption is declarative.
Description of urinary marker of alcohol consumption. | Every 3 months during 1 year
  Urinary Ethylglucuronid (sensitiviy of 62-89% and specificity of 93-99% for alcohol absoption within 30 to 80 hours before urinary test.)
Description of blood marker of alcohol consumption. | Every 3 months during 1 year
  Blood phosphatidylethanol (sensitivity of 90-99% and specificity of 100% for alcohol absorption within 2 to 6 weeks before blood test.)

CONTACTS AND LOCATIONS:
Overall Officials: Helene Donnadieu, MH PD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Department of hepato-gastroenterology and liver transplantation, Montpellier, Occitanie, France